CLINICAL TRIAL: NCT00383201
Title: Long-Term Effect of Multi-Purpose Solutions on Ex-Vivo Wetting Angles of Soft Contact Lenses
Brief Title: Effect of Multi-Purpose Solutions on Ex-Vivo Wetting Angles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-01
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2006-09

CONDITIONS: Contact Lens Care
Keywords: Contact Lens Care

INTERVENTIONS:
Device: OptiFree Multi-Purpose Disinfecting Solution

SUMMARY:
To clinically evaluate the effect of a new multi-purpose disinfecting solution compared to a marketed multi-purpose solution on wettability of soft contact lenses worn for 30 days.

ELIGIBILITY:
* Successful daily wear of FDA Group I or IV soft contact lenses for at least one week.
* Vision correctable to 20/30.
* Normal eyes - no current ocular abnormalities that prevent successful contact lens wear.
* No corneal surgery within the past 12 months.
* No systemic disease that affects that eye or that could be worsened by the use of contact lenses or solutions.
* No over-the-counter or prescription ocular medication.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Efficacy:
Contact lens wetting angle measured ex-vivo
Safety:
Slit-lamp Findings: Eyelids and Conjunctiva; Cornea; Iris, Anterior Chamber
Visual Acuity (Snellen)
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Napier, Study Director — Alcon Research
Locations (1):
- Fort Worth Site, Fort Worth, Texas, United States